CLINICAL TRIAL: NCT01273220
Title: National Epidemiologic Survey on Alcohol and Related Conditions -III
Brief Title: National Epidemiologic Survey on Alcohol and Related Conditions-III
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911056; 11-AA-N056
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Alcohol-Related Disorders
Keywords: Epidemiology; Epidemiologic Survey; Alcohol
MeSH Terms: conditions — Alcohol-Related Disorders

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

- Alcohol use disorders are the most prevalent mental disorders in the United States and are a factor in more than 10 percent of all deaths, including heart disease, stroke, and certain types of cancer and chronic illness. Research into better treatment methods for alcohol use disorders and their associated disabilities requires a broad amount of information on the genetic and environmental factors that predispose certain individuals to alcoholism. To improve the quality of available information for research, the National Institutes of Health is conducting a nationwide survey on alcohol use disorders and related physical and mental disabilities, and will collect genetic information through saliva samples.

Objectives:

- To collect interview data and saliva samples from the U.S. civilian noninstitutionalized population, 18 years and older, in order to study the extent of and contributing factors to alcohol use and abuse in the United States.

Eligibility:

- Individuals at least 18 years of age who do not live in institutions (i.e., prisons, inpatient mental hospitals) and who are willing to be interviewed in English, Spanish, and the four most commonly spoken Asian languages in the United States (e.g., Chinese, Korean).

Design:

* The study will involve three main components: an automated computer-assisted interview, an automated questionnaire, and the collection of a saliva sample.
* Participants will be recruited through community through publically available U.S. Census Bureau files.
* The interview and questionnaire will ask standardized questions related to personal history; alcohol use and possible disorders; symptoms scales of mood, anxiety, and eating conditions that frequently co-occur with alcohol and drug use disorders; tobacco, medicine and drug use and disorders; selected personality traits, including behavior; alcohol, drug, and mental health treatment utilization; and medical conditions related to alcohol consumption.
* Participants will provide a saliva sample for genetic study.

Background:

- Alcohol use disorders are the most prevalent mental disorders in the United States and are a factor in more than 10 percent of all deaths, including heart disease, stroke, and certain types of cancer and chronic illness. Research into better treatment methods for alcohol use disorders and their associated disabilities requires a broad amount of information on the genetic and environmental factors that predispose certain individuals to alcoholism. To improve the quality of available information for research, the National Institutes of Health is conducting a nationwide survey on alcohol use disorders and related physical and mental disabilities, and will collect genetic information through saliva samples.

Objectives:

- To collect interview data and saliva samples from the U.S. civilian noninstitutionalized population, 18 years and older, in order to study the extent of and contributing factors to alcohol use and abuse in the United States.

Eligibility:

- Individuals at least 18 years of age who do not live in institutions (i.e., prisons, inpatient mental hospitals) and who are willing to be interviewed in English, Spanish, and the four most commonly spoken Asian languages in the United States (e.g., Chinese, Korean).

Design:

* The study will involve three main components: an automated computer-assisted interview, an automated questionnaire, and the collection of a saliva sample.
* Participants will be recruited through community through publically available U.S. Census Bureau files.
* The interview and questionnaire will ask standardized questions related to personal history; alcohol use and possible disorders; symptoms scales of mood, anxiety, and eating conditions that frequently co-occur with alcohol and drug use disorders; tobacco, medicine and drug use and disorders; selected personality traits, including behavior; alcohol, drug, and mental health treatment utilization; and medical conditions related to alcohol consumption.
* Participants will provide a saliva sample for genetic study.

DETAILED DESCRIPTION:
The National Epidemiologic Survey on Alcohol and Related Conditions-III (NESARC-III) is planned to be fielded in 2012 by the National Institute on Alcohol Abuse and Alcoholism (NIAAA) in conjunction with Westat, through a contract under data collection authority Title 42 U.S.C. 285 n (Attachment 23.a). The target population of the NESARC-III is the civilian noninstitutionalized population, 18 years and older, residing in the contiguous United States (U.S.) and Alaska and Hawaii. The sample (N=46,500) will include households and selected noninstitutionalized group quarters (e.g., agricultural, vocational training and other dormitories, halfway houses, hostels, YMCAs, shelters, campgrounds, carnivals). The NESARC-III will collect information on alcohol use disorders and related physical and mental disabilities in addition to DNA to be obtained through saliva samples.

This request for IRB approval also includes a pilot test of approximately 50 respondents that will serve the sole purpose of testing the data collection procedures, operations and system architecture of the NESARC-III survey. There will also be two small methodological subcomponents of the NESARC-III proper that will serve the purposes of providing ongoing validation and assessment of the utility of outcome measures appearing on the major data collection questionnaire, the Alcohol Use Disorder and Associated Disabilities Interview Schedule-V (AUDADIS-V: Grant et al., 2008). In the first methodological subcomponent, 1000 respondents participating in the NESARC-III proper will be re-interviewed with a shorter version of the original AUDADIS-V. In the second methodological subcomponent, 700 different respondents participating in the NESARC-III proper will be re-interviewed using a different assessment instrument, the Psychiatric Research Interview for Substance and Mental Disorders (PRISM: Hasin et al., 2008), covering information on major outcome variables very similar to those appearing in the AUDADIS-V. NIAAA has conducted such validation/utility tests that have received OMB approval (OMB No. 0930-0151, OMB No. 0925-0455: Grant et al., 2003a; Ruan et al., 2008) in the past. The design and procedures associated with each of these methodological subcomponents will be explicated and discussed within the body of this IRB submission as necessary.

The NESARC-III will be the fourth national survey conducted by NIAAA. The objectives and content areas of the NESARC-III are extremely similar to those of the prior three NIAAA surveys, with the exception of the NESARC-III s provision for collecting saliva samples. Prior NIAAA national surveys included the 1991-1992 National Longitudinal Alcohol Epidemiologic Survey (OMB No. 0930-0151: Grant et al., 1994), the 2001-2002 Wave 1 NESARC (OMB No. 0925-0484: Grant et al., 2003b), and the 2004-2005 Wave 2 NESARC (OMB No. 0925-0484: Grant et al., 2006).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults, 18 years and older.
* Noninstitutionalized U.S. civilian population living in households.

Selected noninstitutional group quarters including, vocational training and other dormitories, halfway houses, hostels, YMCAs, shelters, campgrounds, carnivals.

-Persons who prefer to have their interviews conducted in English, Spanish, and the four most commonly spoken Asian languages in the U.S.

EXCLUSION CRITERIA:

* Children and adolescents 17 years and younger.
* Military living off base.
* Institutional group quarters including: military living on base, prisons and other correctional facilities; hospitals; nursing homes; hospices; schools; homes or wards for physically handicapped; all juvenile institutions; residential treatment for emotionally disturbed; and homes for abused, dependent and neglected children.
* Persons who prefer to have their interviews conducted in languages other than English, Spanish or the four Asian languages most commonly spoken in the U.S.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36309 (Actual)
Dates: Start 2011-01-07 (Actual); Primary Completion 2013-09-26 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
The prevalence of alcohol and drug use practices
Alcohol and drug use disorders

CONTACTS AND LOCATIONS:
Overall Officials: Tulshi D Saha, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institute on Alcohol Abuse and Alcoholism (NIAAA), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hasin DS, Stinson FS, Ogburn E, Grant BF. Prevalence, correlates, disability, and comorbidity of DSM-IV alcohol abuse and dependence in the United States: results from the National Epidemiologic Survey on Alcohol and Related Conditions. Arch Gen Psychiatry. 2007 Jul;64(7):830-42. doi: 10.1001/archpsyc.64.7.830. PMID 17606817
- [Background] Grant BF, Dawson DA, Stinson FS, Chou PS, Kay W, Pickering R. The Alcohol Use Disorder and Associated Disabilities Interview Schedule-IV (AUDADIS-IV): reliability of alcohol consumption, tobacco use, family history of depression and psychiatric diagnostic modules in a general population sample. Drug Alcohol Depend. 2003 Jul 20;71(1):7-16. doi: 10.1016/s0376-8716(03)00070-x. PMID 12821201
- [Background] Ruan WJ, Goldstein RB, Chou SP, Smith SM, Saha TD, Pickering RP, Dawson DA, Huang B, Stinson FS, Grant BF. The alcohol use disorder and associated disabilities interview schedule-IV (AUDADIS-IV): reliability of new psychiatric diagnostic modules and risk factors in a general population sample. Drug Alcohol Depend. 2008 Jan 1;92(1-3):27-36. doi: 10.1016/j.drugalcdep.2007.06.001. Epub 2007 Aug 13. PMID 17706375